CLINICAL TRIAL: NCT03921034
Title: Pain After Total Knee Arthroplasty: a Comparison of Combined Continuous Adductor Canal Block With Infiltration of Local Anesthetic Between the Popliteal Artery and Capsule of the Knee Block Versus Continuous Adductor Canal Block Alone on Postoperative Analgesia
Brief Title: IPACK Nerve Block for Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Matthew Patterson, Principal Investigator, Ochsner Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016.307.C
Record Dates: First submitted 2019-04-10; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Arthropathy of Knee; Anesthesia
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Only the regional anesthesiologist performing the block will know the randomization status. The study participants, outcome assessors/researchers, other anesthesia personnel, surgeons, physician assistants, and nurses will be blinded to the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuous ACB with IPACK block (Active Comparator): ACB bolused with 20 ml of ropivacaine 0.25% with 1:300,000 epinephrine followed by an 8 ml/hr continuous infusion of ropivacaine 0.2% and IPACK block with 20 ml of ropivacaine 0.25% with 1:300,000 epinephrine
  Interventions: Drug: Ropivacaine
- continuous ACB with sham subcutaneous saline injection (Sham Comparator): ACB bolused with 20 ml of ropivacaine 0.25% with 1:300,000 epinephrine followed by an 8 ml/hr continuous infusion of ropivacaine 0.2% and a sham IPACK block with subcutaneous saline injection along the medial thigh
  Interventions: Drug: Ropivacaine; Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — All patients will receive sedation with midazolam and/or fentanyl titrated to comfort during block procedures. Per our standard practice at Ochsner Medical Center, all patients will have either spinal or combined spinal-epidural anesthesia with mepivacaine 1.5% as the primary anesthetic during the surgery and sedation with propofol titrated to comfort. Also per our standard practice at Ochsner Medical Center, multimodal therapy will include ketamine 0.25mg/kg IV (up to 50mg) intraoperatively, dexamethasone 8mg IV intraoperatively, pregablin 150mg PO preoperatively (adjusted to 75mg for age over 70) followed by 75mg nightly (or home gabapentin dose), acetaminophen 1000mg IV followed by 100mg PO every 6 hours postoperatively, and celecoxib 400mg PO on POD #0 followed by 200mg PO daily.
  Other Names: Naropin
Drug: Saline — All patients will receive sedation with midazolam and/or fentanyl titrated to comfort during block procedures. Per our standard practice at Ochsner Medical Center, all patients will have either spinal or combined spinal-epidural anesthesia with mepivacaine 1.5% as the primary anesthetic during the surgery and sedation with propofol titrated to comfort. Also per our standard practice at Ochsner Medical Center, multimodal therapy will include ketamine 0.25mg/kg IV (up to 50mg) intraoperatively, dexamethasone 8mg IV intraoperatively, pregablin 150mg PO preoperatively (adjusted to 75mg for age over 70) followed by 75mg nightly (or home gabapentin dose), acetaminophen 1000mg IV followed by 100mg PO every 6 hours postoperatively, and celecoxib 400mg PO on POD #0 followed by 200mg PO daily.
  Arms: continuous ACB with sham subcutaneous saline injection

SUMMARY:
Double-blind, randomized controlled clinical trial to test the efficacy of IPACK on postoperative opioid consumption, patient satisfaction, pain scores, mobility, and several other secondary outcomes in adults undergoing primary unilateral TKA.

Enrolled patients will be randomized to either continuous ACB with IPACK or to continuous ACB with sham subcutaneous saline injection. Outcomes assessors and patients will be blinded to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral, primary tricompartment total knee arthroplasty
* Age 18 years or older
* ASA I-III
* Eligible for spinal or combined spinal epidural anesthetic
* Able to speak, read, and understand English
* Willing to participate in the trial

Exclusion Criteria:

* Contraindication to regional anesthesia or peripheral nerve blocks
* Allergy to local anesthetics
* Allergy to NSAIDs
* Chronic renal insufficiency with Cr > 1.4 or GFR < 60
* Have chronic pain that is not related to their knee joint
* Have been using opioids on a chronic basis (daily or almost daily opioid use for 3 months or longer)
* Have a pre-existing peripheral neuropathy involving the operative site
* Body mass index greater than or equal to 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption (morphine equivalents) in the first 24 hours | 24 hours

SECONDARY OUTCOMES:
Patient satisfaction on day of discharge using the Brief Pain Inventory (BPI) or a similar validated satisfaction survey | through study completion approximately 2 days
Average pain score at rest and with physical therapy in PACU, POD#1 am, POD#1 pm | through study completion approximately 2 days
Worst pain score at rest and with physical therapy in PACU, POD#1 am, POD#1 pm | through study completion approximately 2 days
Walk distance on POD#1 am, POD#1 pm, POD#2 | through study completion approximately 2 days
Time to first intravenous opioid, oral opioid in PACU and after arrival to hospital room | through study completion approximately 2 days
Time to oral-only opioids | through study completion approximately 2 days
Pain location | through study completion approximately 2 days
Hospital length of stay | through study completion approximately 2 days
Incidence of foot drop | through study completion approximately 2 days
Incidence of itching, nausea, or vomiting in PACU, POD#1am, POD#1 pm | through study completion approximately 2 days
Incidence of over-sedation based on Richmond Agitation Sedation (RASS) score | through study completion approximately 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Patterson, MD, Principal Investigator — Ochsner

IPD SHARING:
Plan to Share IPD: No
No plan

DOCUMENTS (2):
  • Informed Consent Form (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT03921034/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT03921034/Prot_SAP_001.pdf